CLINICAL TRIAL: NCT00365118
Title: Treatment of Naevus Flammeus Using Intense Pulsed Light and Pulsed Dye Laser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: KF-01-278867
Record Dates: First submitted 2006-08-15; First posted 2006-08-17 (Estimated); Last update posted 2008-06-03 (Estimated); Status verified 2008-06

CONDITIONS: Port-Wine Stain
Keywords: Port wine stains; naevus flammeus
MeSH Terms: conditions — Port-Wine Stain; Hemangioma, Capillary | interventions — Lasers, Dye

INTERVENTIONS:
Device: Pulsed dye laser (Candela), Intense pulsed light (Palomar)

SUMMARY:
The purpose of the trial is to compare efficacy and adverse effects of pulsed dye laser and intense pulsed light in patients with port wine stains.

ELIGIBILITY:
Inclusion Criteria:

* Patients with previously untreated and previously laser-treated naevus flammeus. Naevus flammeus measuring at least 5 x 7 cm within a single anatomical area. For example, the face corresponding to dermatomes V1, V2 and V3, back, abdomen, arms and legs.Patients aged two or above.Patients with skin types I-III.

Exclusion Criteria:

* Patients below two years of age.
* Pregnant or breastfeeding patients.
* Patients with known increased sensitivity to visible light.
* Patients with a tendency to produce hypertrophic scars or celoids.
* Patients with skin types IV, V and VI.
* Patients who are clearly pigmented following recent exposure to the sun or a solarium.
* Patients treated with Roaccutane during the last six months.
* Patients who are not considered able to follow the treatment protocol (e.g. severely alcoholic patients, dementia patients, mentally ill patients, etc.).

Min Age: 2 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Dates: Start 2005-11; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merete Hædersdal, MD, PhD, DrMedSci, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen, Copenhagen Nv, Denmark